CLINICAL TRIAL: NCT05888987
Title: Use of a New Rapid Multiplex PCR System for the Microbiological Diagnosis of Severe Infectious Keratitis: Impact on Therapeutic Management (ABCORFILM Study)
Brief Title: Use of a New Method for the Microbiological Diagnosis of Severe Corneal Infection
Acronym: ABCORFILM
Status: Recruiting | Type: Observational
Sponsor: CHU de Reims (Other)
Responsible Party: Sponsor
Other Study IDs: PA23064
Record Dates: First submitted 2023-05-25; First posted 2023-06-05 (Actual); Last update posted 2024-09-19 (Actual); Status verified 2024-09

CONDITIONS: Infectious Keratitis; Microbial Keratitis; Corneal Infection
Keywords: Severe infectious keratitis; Infectious keratitis; Microbial keratitis; Corneal infection; FilmArray; Multiplex PCR system

STUDY DESIGN:
Observational Model: Other | Time Perspective: Other
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Before
- After
  Interventions: Biological: PCR multiplex by FilmArray

INTERVENTIONS:
Biological: PCR multiplex by FilmArray — PCR multiplex by FilmArray system on corneal swabbing sample
  Groups: After

SUMMARY:
Microbial keratitis is a severe and often blindness-inducing pathology which represents today the first reason for long-term hospitalization (more than 5 days) in ophthalmology. Its diagnosis is clinical and leads to an immediate hospitalization in the presence of serious criteria (Mackie classification). The entire process of microbiological diagnosis requires several days before etiological confirmation and therefore delays the initiation of targeted therapy.

Recently, new PCR systems allowing the detection of 18 to 27 pathogens in 75 minutes have been developed. Their use could thus be transposed to ophthalmology by adapting the microbiological diagnostic technique to samples currently taken by swabbing the cornea.

The investigators will compare their diagnosis performance versus conventional methods on patients who suffered for a microbial keratitis with severity criteria.

DETAILED DESCRIPTION:
46 patients enrolled for severe infectious keratitis will be recruited in the department of Ophthalmology, Robert Debré Hospital, Reims, France. The study will be composed by 2 groups. The first, also called "before group" will contain 23 patients who were anteriorly hospitalized for a severe infectious keratitis in our hospital unit. They received standard microbiological diagnosis methods: Direct microscopic examination with Gram stain, bacterial and fungal cultures, viral and amoebic polymerase chain reaction [PCR]).

The second, also called "after group" will enroll patients who suffer for a severe infectious keratitis (prospective group). Each patient will benefit a complete ophthalmologic examination, corneal scrapping and swabbing for standard microbiological diagnosis methods along with another corneal swabbing sample for the use of two different FilmArray® PCR systems identified as "ME" for Meningitis-Encephalitis and "BCID" for Blood Culture Identification.

The investigators hypothesize that the use of rapid multiplex PCR tests for the microbiological diagnosis of severe corneal infections could in the future prove to be more efficient than the current diagnostic strategy, on the one hand, by shortening the time to identify the pathogen and therefore to implement a targeted treatment, and on the other hand, by systematically searching for a large number of pathogens well beyond those targeted today. In addition, the benefits of this technique applied to ophthalmology could improve the long-term visual prognosis, reduce the length of hospitalization and therefore the diagnostic and management costs of these patients.

ELIGIBILITY:
Inclusion criteria:

* Over 18 years old
* With social security affiliation
* Willing to participate this study
* Hospitalized in our department for severe infectious keratitis

Non-inclusion criteria:

* Any prior (48 hours) or concomitant treatment with local or systemic antibiotherapy at time of corneal scrapping and swabbing
* Patient not covered by the French Health Insurance
* Unable to give informed consent

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Adult patients treated for a severe corneal abscess according to the Mackie classification (requiring hospitalization) at the Reims University Hospital between 05/01/2022 and 04/30/2023 ("before" phase) and between 01/ 05/2023 and 04/30/2024 ("after" phase).
Sampling Method: Non-Probability Sample
Enrollment: 46 (Estimated)
Dates: Start 2023-07-07 (Actual); Primary Completion 2027-01-07 (Estimated); Study Completion 2027-08-07 (Estimated)

PRIMARY OUTCOMES:
Time to modification of the first line antimicrobial treatment towards a treatment targeting the detected pathogen. | At 2 weeks

SECONDARY OUTCOMES:
Duration of hospitalization | At 1 month
Best corrected visual acuity | At 12 months
Modification of the initial antimicrobial treatment after detection of the etiological agent | At 1 month
Descriptive analysis of pathogens responsible for severe infectious keratitis in Champagne-Ardenne | At 1 month
• Costs of diagnostic methods (conventional and FilmArray) and management (cost of the average length of stay in ophthalmology at the Reims University Hospital for severe infectious keratitis) | At 1 month

CONTACTS AND LOCATIONS:
Locations (1):
- Damien JOLLY, Reims, France